# **Dietary Nitrate and Muscle Power with Aging**

Principal Investigator: Andrew Coggan, Ph.D.

Associate Professor, Department of Kinesiology I.U. School of Health and Human Sciences

Sub-Investigators: Ranjani N. Moorthi, M.D.

Sharon Moe, M.D. Tarah Ballinger, M.D. Ziyue Liu, Ph.D. Edgar Gallardo

# **Table of Contents:**

# **Study Schema**

- 1.0 Background
- 2.0 Rationale and Specific Aims
- 3.0 Inclusion/Exclusion Criteria
- 4.0 Enrollment/Randomization
- **5.0** Study Procedures
- **6.0** Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others
- 7.0 Study Withdrawal/Discontinuation
- 8.0 Statistical Considerations
- 9.0 Privacy/Confidentiality Issues
- 10.0 Follow-up and Record Retention
- 11.0 References
- 12.0 Appendix

## 1.0 Background

Aging is accompanied by a progressive reduction in the maximal strength, speed, and especially <u>power</u> of skeletal muscle. These age-related physiological changes often lead to functional limitations that are highly predictive of disability, institutionalization, and mortality in the elderly (1,2). Thus, <u>any intervention that significantly enhances muscle contractile properties could potentially improve the health, quality of life, and possibly even the longevity of older individuals.</u>

Numerous factors undoubtedly account for the decline in muscle function, with agerelated changes in the size, properties, and neural control of muscle likely all playing a role (3). Another important factor, however, may be a fall in nitric oxide (NO) bioavailability with aging. Although initially identified as a vasodilator, i.e., as "endothelium-derived relaxing factor", NO is in fact a key cellular signaling molecule with pleiotropic effects in many tissues. These include skeletal muscle, wherein among other effects NO helps modulate contractile function (cf. Refs. 4-8 for review). Specifically, during *isometric* contractions NO may, or may not, slightly suppress maximal force production (4-8). This may be due to nitrosation or S-nitrosylation of various proteins (9). During *concentric* activity, however, NO significantly increases the rate of force development, maximal shortening velocity, and maximal *power* of both single muscle fibers and isolated muscles (4-8).

Based on animal studies, these stimulatory effects are thought to be mediated via activation of the classic NO-sGC-cGMP pathway (10), and have been *euphemistically* described by Maréchal and Gailly (5) as a "slow-to-fast" shift *qualitatively* akin to the chronic transformation of muscle fiber type that occurs with, e.g., prolonged electrical stimulation. With aging, however, whole-body NO production decreases, as evidenced, e.g., by a progressive decline in the plasma concentrations of its downstream metabolites,  $NO_2^-$  and  $NO_3^-$  (11,12). In skeletal muscle itself, there is a dramatic decrease in interstitial  $NO_2^-$  and  $NO_3^-$  concentrations (13), as well as a reduction in intracellular  $NO_3^-$  content (14) These changes are accompanied by a decline in the activity of the neuronal form of NO synthase (nNOS, or NOS1) (15,16), the primary isoenzyme within muscle responsible for the synthesis of NO from L-arginine,  $O_2$ , and NADPH. This is associated with an age-related reduction in flow-mediated vasodilation



Figure 1. NO-sGC-cGMP signaling via the enterosalivary. From Ref. 22.

(17-20), perhaps the hallmark indicator of NO bioavailability. In turn, the latter (i.e., flow-mediated vasodilation) has been shown to correlate positively with muscular power and physical functioning in older men and women (21). Taken together, these data suggest that decreased skeletal muscle NO production may contribute to the age-associated decline in muscle contractile properties and hence in functional capacity.

In this context, the physiological effects of dietary NO<sub>3</sub><sup>-</sup> are of considerable interest. It

is now recognized that  $NO_3$  in the diet is a significant source of NO in body (22-26) (**Fig. 1**).

In fact, this dietary pathway, which entails the reduction of  $NO_3^-$  to  $NO_2^-$  by facultative anaerobic bacteria in the mouth followed by further reduction of  $NO_2^-$  to NO by, e.g., deoxyhemoglobin, can account for up to ~25% of basal whole-body NO production (27,28). This dietary pathway serves as an important "backup" system to the more well-known NOS pathway. This is likely to be especially true in skeletal muscle, since unlike the NOS pathway the dietary pathway operates well at low  $pO_2$  and is stimulated rather than inhibited by low pH (22-26), conditions that regularly exist in muscle, both at rest and especially during contractile activity. Indeed, skeletal muscle has recently been shown to play a central role in  $NO_3^-/NO_2^-/NO$  metabolism (29).

Haider and Folland (30) and Whitfield et al. (31) have reported that dietary NO<sub>3</sub><sup>-</sup> intake enhances the rate of force development and peak force output of the human quadriceps muscle during electrically-stimulated contractions. Numerous recent studies (reviewed in 32) demonstrate that dietary NO<sub>3</sub><sup>-</sup> can enhance other types of exercise performance in various subject groups. To date, however, only a handful of studies have specifically examined the impact of dietary NO<sub>3</sub><sup>-</sup> on exercise capacity in older individuals (33-35). These studies found no effect of consuming 9.6-12 mmol NO<sub>3</sub>-/d for 3-7 days on various measures of aerobic exercise performance in healthy older men and women (33,34) or in older individuals with hypertension or heart failure (HF) (35). Similarly, Justice et al. (36) reported that ingesting NO<sub>2</sub> (not NO<sub>3</sub>) at 1.2-2.4 mmol/d for 10 weeks did not improve VO₂max in middle-aged and older study participant, although it did increase the rate of force development (but not maximal force, i.e., strength) during isometric muscle contractions. Importantly, however, *none* of these studies of older study participant measured maximal muscle power. The effects of dietary NO<sub>3</sub>- on this critical aspect of muscle contractile function in older study participant are therefore still completely unknown. Moreover, it cannot be automatically assumed that dietary NO<sub>3</sub> will be equally efficacious in improving muscle function in older persons as we have found in other study participant groups (37-39). For example, in rodents, the effects of dietary NO<sub>3</sub> are more prominent in fast- vs. slow-twitch muscle (40,41), and some (42-45), but not all (46-48), studies of humans have found that aging results in a reduction in the percentage of fast-twitch muscle fibers. Alternatively and/or in addition, more rapid destruction of NO due to increased production of reactive oxygen species by aging muscle (49) could limit the beneficial effects of dietary NO<sub>3</sub><sup>-</sup> on muscle NO-sGC-cGMP signaling in older persons

Even if it can be shown that dietary  $NO_3^-$  acutely improves muscle function in older men and women, it remains to be established whether such benefits can be sustained, and/or whether such effects have a positive impact on a person's daily life. This is not necessarily a given, as it is well known that tolerance develops quite quickly in response to *pharmacological* nitrates, e.g., glyceryl trinitate (nitroglycerin) (49). This does not seem to be true, though, for dietary  $NO_3^-$  (50,51) – in fact, animal studies indicate that ingestion of  $NO_3^-$  for 5-7 days may lead to positive adaptations in calcium handling proteins and hence force production in muscle that would tend to mitigate age-related declines in these parameters (40). Notably, however, a recent study of humans was unable to reproduce these findings (31).

Our **Preliminary Data** suggest that the effects of dietary  $NO_3^-$  on muscle speed and power are maintained (but not enhanced) for at least 14 days with <u>repeated</u> (i.e., daily) dosing in humans (see below).

#### Preliminary data

Using methods essentially identical to those to be employed in the proposed experiments, including use of a "gold standard", double-blind, placebo-controlled, crossover design, we previously demonstrated that dietary  $NO_3^-$  intake increased maximal knee extensor speed (Vmax) and power (Pmax) in 12 healthy, younger men and women by  $11\pm5\%$  (P<0.05) and  $6\pm3\%$  (P<0.05), respectively (37). We observed similar dietary  $NO_3^-$ -induced improvements in muscle speed and power in 13 athletes performing multi-joint, multi-muscle, i.e., sprint cycling, exercise (38). Lastly, we found even greater increases in Vmax and Pmax (of  $12\pm5\%$ , P=0.09, and  $13\pm4\%$ , P<0.05, respectively) in nine middle-aged patients with systolic heart failure (HF) (52). The greater beneficial effect of dietary  $NO_3^-$  in HF patients presumably reflects the fact that, similar to healthy aging, HF results in reduced NO bioavailability (53).

Using the same methods, we have also recently determined the effects of acute dietary  $NO_3^-$  intake in seven men and women 61-78 y of age. As shown in **Table 1**, plasma  $NO_3^-$  and  $NO_2^-$  and breath NO increased (P<0.05) by  $1309\pm188\%$ ,  $268\pm91\%$ , and  $146\pm19\%$ , respectively, by 2 hours after ingestion, and all three remained elevated for the remainder of the experiment. These observations are consistent with previous research in older study participant demonstrating that plasma  $NO_3^-$  and  $NO_2^-$  concentrations peak 2-3 hours after ingestion of a  $NO_3^-$  load (54), which is comparable to the time course observed in younger study participant (55-57).

Table 1. Changes in plasma  $NO_3^-$  and  $NO_2^-$  and breath NO in response to dietary  $NO_3^-$  intake in older study participant.

| | <u>Trial</u> | <u>Pre</u> | <u>1 h</u> | <u>2 h</u> | 10 min post exer. |
|---|---|---|---|---|---|
| Plasma NO <sub>3</sub> - (µmol/L) | Placebo | 26±4 | 24±3 | 24±3 | 22±4 |
| | Nitrate | 31±7 | 285±27* | 295±27* | 282±33* |
| Plasma NO <sub>2</sub> - (µmol/L) | Placebo | 0.21±0.03 | $0.26 \pm 0.06$ | $0.26 \pm 0.06$ | $0.20\pm0.03$ |
| | Nitrate | 0.27±0.04 | $0.43 \pm 0.13$ | 0.49±0.06* | 0.56±0.10* |
| Breath NO (ppb) | Placebo | 23±5 | 26±4 | 27±4 | 23±5 |
| | Nitrate | 27±4 | 49±7* | 38±4* | 52±10* |

Values are mean  $\pm$  S.E. for n=7. \*Nitrate trial significantly higher than Placebo trial at same time point (P<0.05).

Fig. 2 Changes in maximal knee extensor speed (Vmax, top panel) and power (Pmax; bottom panel\_ in response to dietary NO<sub>3</sub>-; intake in older adults



As shown in **Fig. 2**, dietary  $NO_3^-$  intake increased Vmax in six out of seven of these study participants, with the average improvement being  $9\pm3\%$  (P<0.05). Pmax

increased in five out of the seven study participants, with the average increase being  $4\pm3\%$  (P=0.15). These preliminary results, which were presented at the  $64^{th}$  annual American College of Sports Medicine meeting in Denver, CO, May 30-June 3, 2017, are similar to those we obtained previously in younger individuals (37), and thus support our primary hypothesis.

Biopsy samples were obtained from the v. lateralis of two of these study participant  $\sim 3$  h after ingestion of either the placebo or  $NO_3^-$  and analyzed for cGMP content. As shown in **Fig. 3**, muscle cGMP was higher in both study participants in the  $NO_3^-$ 





Figure 3. Effect of NO<sub>3</sub> ingestion on muscle cGMP content.

Another of the study participants (number 5) continued to ingest either the NO<sub>3</sub><sup>-</sup> supplement or the placebo daily for a total of 14 days, separated by a 10 day washout period. As shown in **Fig. 4**, their Pmax and Vmax were

enhanced almost identically after both acute and chronic ingestion, such that the two dashed curves are superimposable. These data demonstrate that tolerance does not develop in response to repeated ingestion of dietary NO<sub>3</sub><sup>-</sup>. Furthermore, since Vmax and Pmax were comparable after 14 vs. 1 day of placebo treatment (i.e., 25 vs. 11 day post NO<sub>3</sub><sup>-</sup> treatment), they also indicate that even a 10 day washout period (vs. the 14 days we propose to use) is sufficient to eliminate any carryover effects.

In summary, we have demonstrated that dietary NO<sub>3</sub><sup>-</sup> improves maximal muscle speed and power in a variety of subject populations, including a small number of healthy, elderly men and women. Furthermore, we have demonstrated that dietary NO<sub>3</sub><sup>-</sup> intake results in an increase in muscle NO-sGC-cGMP signaling. Finally, we have demonstrated that daily ingestion of dietary NO<sub>3</sub><sup>-</sup> for 14 days does not result in tolerance. These preliminary data therefore provide very strong support for the current study.



Figure 4. Effects of acute vs. chronic dietary NO<sub>3</sub>- intake on maximal knee extensor power (Pmax) and speed (Vmax) in a 78 y old woman.

## 2.0 Rationale and Specific Aims

We hypothesize that increased dietary NO<sub>3</sub> intake will enhance muscle NO-sGC-cGMP signaling in older men and women, leading to an increase in maximal speed and power.

Helping drive our hypotheses are the consistent improvements in muscle speed and power that both we and others have observed following dietary NO<sub>3</sub><sup>-</sup> intake in healthy younger study participants (37), athletes (38,39), and especially heart failure patients (52).

By focusing specifically on changes in muscle contractile properties, we will not be able to determine whether dietary  $NO_3^-$  supplementation reduces the  $O_2$  cost of exercise in older study participant. We will also not be measuring the effect of acute and/or chronic dietary  $NO_3^-$  intake on muscle blood flow, or on muscle energetics or aerobic exercise performance. We will also not be testing whether dietary  $NO_3^-$  intake improves insulin sensitivity. In preliminary experiments, however, we have not been able to reproduce the  $O_2$ -sparing effect of  $NO_3^-$  ingestion, and several recent studies have reported that dietary  $NO_3^-$  (or  $NO_2^-$ ) does not significantly improve aerobic exercise function in older men and women (32-35). Similarly, several other recent studies have demonstrated that, contrary to the results of *in vitro* or animal experiments, dietary  $NO_3^-$  does not enhance insulin sensitivity in older humans (58-60). We therefore believe that we are well-justified in focusing on changes in muscle contractile properties, especially in light of our preliminary data and the important role that reductions in muscle function play in the aging process.

Because our focus is muscle contractile function, we considered using percutaneous electrical nerve stimulation rather than voluntary exercise. However, this approach inverts the normal orderly recruitment of motor units, preferentially depolarizing larger alpha motor neurons innervating type II muscle fibers (cf. 61 for review). Thus, while potentially magnifying the effects of dietary  $NO_3^-$  on muscle speed and power it would significantly diminish the external validity of our findings.

We considered, but rejected, various alternatives to our "gold standard", double-blind, placebo-controlled, crossover design. This design is the most efficient for testing all of our hypotheses, i.e., it requires the fewest number of study participant to provide adequate statistical power (since each subject serves as their own control). A cross-sectional study would require >10x study participant to provide equivalent power for detecting changes in Pmax.

Finally, we note that historically there have been concerns that increased  $NO_3^-$  intake may lead to formation of carcinogenic nitrosamines (62). However, the Joint FAO/WHO Expert Committee on Food Additives has concluded that "Overall, the epidemiological studies showed no consistently increased risk for cancer with increasing consumption of  $NO_3^-$ ." (63). Furthermore, diets high in vegetables, such as the DASH diet widely recommended to hypertensive patients, routinely exceed the WHO acceptable daily intake of  $NO_3^-$  by >5-fold. In contrast, the amount of dietary  $NO_3^-$  shown to improve exercise tolerance in previous studies is only slightly above the WHO limit (63). Nonetheless, the safety and efficacy of increased dietary  $NO_3^-$  would need to be established in follow-up large-scale, longer-term studies before beet root juice (BRJ) or other  $NO_3^-$ -rich foods could be widely recommended to older individuals.

**Specific Aim #1:** Determine the *acute* effects of dietary NO3- intake on

muscle NO-sGC-cGMP signaling and muscle contractile

properties

**Specific Aim #2:** Determine the cumulative or *chronic* effects of dietary

NO3- intake on muscle NO-sGC-cGMP signaling and muscle

contractile properties

**Exploratory Aim #3:** Assess the effects of dietary NO3- supplementation on

perceived fatigue, physical function, and physical activity during daily life via questionnaires and accelerometer data

## 3.0 Inclusion/Exclusion Criteria

#### Inclusion:

- Men and women age 65-79
- In good health, as determined by the physician's review of history, physical examination, EKG, and routine blood tests
- Agrees to also participate in the FIT study (IRB # 1707550885).

#### **Exclusion:**

- Men and women <65 or >79 years of age
- Unable to provide informed consent
- Currently pregnant or lactating
- Current smokers
- Significant orthopedic limitations or other contraindications to strenuous exercise
- Those taking phosphodiesterase inhibitors (e.g., Viagra)
- Those taking proton pump inhibitors, antacids, xanthine oxidase inhibitors, or on hormone replacement therapy
- History of major metabolic disease (e.g., type I and type II diabetes, thyroid disorders), neuromuscular disease (e.g., cervical spondylotic radiculomyelopathy, lumbar spondylosis, amyotrophic lateral sclerosis, Guillain-Barré syndrome, and acquired demyelinating polyneuropathies), cardiovascular disease (e.g., > stage II hypertension, heart failure, myocardial infarction/ischemia, significant myocardial or pericardial diseases (e.g. amyloidosis, constriction), moderate or severe valvular disease, renal disease, liver disease, or anemia
- Expending greater than 1500 kcal/week in moderate or greater intensity physical activity as defined by the CHAMPS physical activity questionnaire

One hundred study participants will be enrolled to attain sixteen completed participants.

## 4.0 Enrollment/Randomization

Subjects will be recruited from the community through approved methods including flyers, emails from the Indiana Clinical and Translational Sciences Institute (All IN for Health), NIH sponsored website/email via ResearchMatch.org and newspaper advertisements.

In addition, our study will be listed on the Indiana CTSI study listing called the All IN for Health TrialX iConnect. iConnect is a HIPAA-compliant and secure public facing research recruitment platform provided by the Indiana Clinical and Translational Sciences Institute (Indiana University) consisting of a study trial listing and volunteer registry. This system is licensed by Indiana University from TrialX and is monitored by the Indiana University Information Technology Services (UITS) and University Information Security Office (ISO). Study Teams have access to their study listings and participant referrals based on a secure login. There is a small Administrative Team within the Indiana CTSI that manages the iConnect platform and has access to all study information, referrals, and registry volunteers. This online platform provides researchers with the ability to create a public facing webpage that can contain a brief prescreener and the ability for the public to refer themselves to the trial: (https://research.indianactsi.org). The study listing information can be modified based on the study and targeted population and provides a direct,

easily managed system to enhance communication with the public. Study teams can also use this webpage as the landing or referral page for any marketing materials that are being used (either by listing the hyperlink or creating a scannable QR code). We have included a screenshot of our study listing for your review and approval. Please see attachment titled "Screenshot iConnect". In addition, potential participants can complete a pre-screener that will determine their preliminary eligiblilty (see attachment "Prescreener for iConnect.")

The study listings are open to the public and any persons who visit our study page may submit their contact information to us through the listing. We can access that information by logging in to our iConnect dashboard. We may respond to and contact interested volunteers directly through the platform or by university phone or email. We will use the following guide for any email responses for phone conversations with the volunteers. For our standard messaging, please see attached "iConnect Study Team Reply Email Message."

In addition to the study listing(s), potential participants will be identified from the Indiana CTSI All IN for Health voluntary registry IU IRB Protocol Number 1105005444. This registry was created so that interested individuals could create a volunteer profile to receive information about ongoing studies. Persons in this registry have provided their self-reported health information for the purposes of being matched to appropriate research studies. The registry volunteers have signed an electronic consent/authorization so that their information can be used and they can be contacted for this reason.

We can also match participants in the registry and are able to send out a message to them through the system in a de-identified manner. We may use the search and filter tool in the system to identify a group of volunteers who match our study criteria based upon the information that the volunteers have included in their profiles. We may then send an outreach message to those de-identified matched volunteers through the online system. If we send an outreach message to matched volunteers, we will use standard messaging (please see attached "iConnect Volunteer Outreach Email Message Template." Matched volunteers who receive our outreach message and indicate they are interested and agree to be contacted specifically for this study will approve for their contact information to be accessible by us through the iConnect portal. If we contact those interested matched volunteers by email or phone, we will use the language from Template C [file name of "iConnect Study Team Reply Email Message" for any email responses for phone conversations with the matched volunteers.

When potential study subjects contact the study team expressing an interest in the study they will be given additional information regarding the study procedures, requirements, and risks. If they are still interested the study team will complete a brief phone screening to see if they qualify for an in-person screening visit. As previously approved by amendment, potential subjects will be asked if they are part of the IU Health medical system and if so, do they give verbal permission for their records to be reviewed for possible exclusions to participation. If they are not part of the IU Health system or do not give permission, they will still be able to participate in a screening visit. If it appears they are eligible for a screening visit, they will be scheduled and a consent form will be mailed / emailed to them ahead of the screening visit for review. After the study participant has had several days to review the consent form, a study team member will call to answer any questions the participant may have regarding the consent form. Subjects will be asked

to fast for 12 hours prior to their screening visit, before they sign the consent form. When the subject arrives for the screening visit, a member of the research team will thoroughly review the consent with the study participant and answer questions. Study participants will be given as much time as they wish to consider participation before signing the consent form. If the study participant agrees to move forward with the screening visit, the consent will be signed by the study participant and the person who reviewed the consent and obtained the participant's signature. A copy of the signed consent form will be provided. Both the participants and the investigators will be blinded to the order of treatment, which will be randomized by the study statistician.

A separate consent form for participation in the Fit Core (IRB study #1707550885) will be administered by the Fit Core staff according to their policies and procedures.

## 5.0 Study Procedures

## Study Design

A diagram of the flow of the study for each participant is shown in **Figure 6.** 



Each participant will be studied using a double-blind, placebo-controlled, crossover design.

The dose of  $NO_3^-$  to be given, which is roughly the equivalent of 3-4 whole beets or 2 cups of cooked spinach (64), has been chosen based on our previous results (37,38,52) and preliminary data, as well as a recent study by Wylie et al. (55) demonstrating that, acutely (i.e., as a single dose), at least 8.4 mmol are needed to elicit an improvement in exercise performance but additional improvement does not result from a dose of 16.8 mmol. The placebo, also to be purchased from James White Drinks Ltd., is prepared by extracting  $NO_3^-$  from beetroot juice (BRJ) using an ion exchange resin and is indistinguishable in packaging, color, taste, texture, and smell from the standard product. Importantly, this placebo does not alter plasma  $NO_3^-/NO_2^-$  or breath  $NO_3^-/NO_2^-$ 

#### Study Procedures

**On Visit 1** (Pre-test), all study participants will complete a screening examination: questionnaires will be completed regarding their physical activity and perceived fatigue and physical function. The participant will undergo a complete history and physical exam by a study physician, an EKG, and phlebotomy for screening and laboratories (complete blood count, liver and kidney function tests, electrolytes, fasting glucose and insulin), and an urine test to assess kidney function. They will also practice the entire

isokinetic dynamometer exercise test. Participants will then be escorted to the Fit Core where Fit Core staff will consent and then complete the Fit Core protocol (IRB study #1707550885).

Participants will be instructed to consume their normal diet (aside from the BRJ supplement) throughout the study. They will, however, be asked to avoid consumption of high  $NO_3^-$  foods (e.g., beets, spinach, collard greens) the evening prior to testing. This approach is justified based on the short half-life of  $NO_3^-$  in plasma (i.e.,  $\sim 8$  hours; Ref. 27) as well as previous research demonstrating that even a *chronic* increase in dietary  $NO_3^-$  intake up to 2.5 mmol/d (i.e.,  $\sim 3x$  normal dietary  $NO_3^-$  intake in the U.S. (54) has no significant influence on plasma  $NO_3^-$  levels (54). Participants will be asked to refrain from using chewing gum, alcohol, and caffeine-containing food/drinks for 24 hours prior to each remaining visit. Participants will also be instructed to refrain from use of an antibacterial mouthwash throughout the study, since this would limit conversion of  $NO_3^-$  to  $NO_2^-$  by bacteria in the oral cavity (65,66). Participants will be asked to fast for 12 hours prior to each remaining study visit.

**On Visit 2** (Day 1 pre-crossover), study participants will complete questionnaires (PROMIS® questionnaire) regarding their perceived fatigue and physical function, will have their vital signs assessed, and will undergo phlebotomy for NO<sub>3</sub><sup>-</sup> and NO<sub>2</sub><sup>-</sup> measurement. They will then ingest 140 mL of BRJ either containing or depleted of 11.2 mmol of NO<sub>3</sub><sup>-</sup> (i.e., **BRJ w/ NO<sub>3</sub>**<sup>-</sup> or **BRJ w/o NO<sub>3</sub>**<sup>-</sup>). After allowing 2 hours for absorption, they will undergo the isokinetic dynamometer. After completion of the dynamometer assessment, subjects will complete the Fit Core protocol, less the DEXA scan. Blood samples will be obtained at hourly intervals during the study. Heart rate and blood pressure will be measured at the same scheduled times as blood samples after which a final blood sample will be obtained. The sequencing of the measurements have been chosen to minimize potential interference/carryover effects that might influence the data and/or its interpretation.

Following completion of the above tests, the participant will continue to ingest 140 mL of BRJ w/  $NO_3^-$  or BRJ w/o  $NO_3^-$  every morning for an additional 13 days, after which the protocol described above will be repeated on the  $14^{th}$  day. To encourage compliance with the experimental protocol and enhance subject retention, the subjects will be initially provided with only a 7 day supply of BRJ. They will also be asked to keep and return the empty BRJ bottles at the next visit.

**On Visit 3** (Day 7 pre-crossover), participants will be asked to return the empty BRJ bottles. At this visit, participants will have their vital signs assessed and a blood sample will be obtained to quantify plasma  $NO_3^-$  and  $NO_2^-$  concentrations. Participants will be asked to rate their perception of fatigue and physical function during the previous week using the NIH-funded Patient-Reported Outcomes Measurement Information System (PROMIS®). The final 7 days of BRJ will be provided. They will also be asked to keep and return the empty BRJ bottles at the next visit.

**On Visit 4** (Day 14 pre-crossover), participants will be asked to return to undergo the same studies as described above for Study Day 2. In addition, participants will be asked to rate their perception of fatigue and physical function during the previous week using the NIH-funded <u>Patient-Reported Outcomes Measurement Information System</u>

(PROMIS®). The study team member will also complete BRJ accountability for the 2<sup>nd</sup>, 7-day consumption period by collecting the empty BRJ bottles

Then the study participant will undergo a 14 day (minimum) washout period consuming neither either **BRJ w/ NO**<sub>3</sub><sup>-</sup> nor **BRJ w/o NO**<sub>3</sub><sup>-</sup>. After this, the study participant will be crossed-over to receive whichever treatment they did not receive first.

**On Visit 5** (Day 1 post-crossover), the study participant will undergo the same procedures as described for Study Day 2.

**On Visit 6** (Day 7 post-crossover), the study participant will undergo the same procedures as described for Study Day 3

**On Visit 7** (Day 14 post-crossover), the study participant will undergo the same procedures as described for Study Day 4.

During each 14 day intervention period (i.e., between Study Days 2 and 4 and 5 and 7 inclusive), an Actigraph wGT3X-BT activity monitor will be worn at the hip during all waking hours except when bathing or swimming. The Actigraph measures ambient light and also accelerations in all three directions, from which total activity counts, active time, sedentary time, sleep, etc., are estimated/quantified.

Subjects will complete a log indicating the times that they wore the activity monitor and return it to the study staff at each visit.

## Study Methods

Measurement of  $NO_3^-$  in each batch of BRJ w/ or w/o  $NO_3^-$ : The  $NO_3^-$  content of each batch of BRJ w/ or w/o  $NO_3^-$  will be determined using high performance liquid chromatography (HPLC) (ENO-30, Eicom USA, San Diego, CA).

Measurement of plasma  $NO_3^-$ ,  $NO_2^-$ : Venous blood samples will be obtained prior to consumption of BRJ w/ or w/o  $NO_3^-$  and every hour thereafter for 3 hours, plasma rapidly separated by centrifugation, and frozen at -80° C until subsequently analyzed for  $NO_3^-$  and  $NO_2^-$  concentration using HPLC as described above.

Measurement of skeletal muscle contractile function: A Biodex 4 system will be used to measure each subject's muscle contractile properties as previously described (30,33). Briefly, study participant will perform maximal knee extensions with their dominant leg at angular velocities of 0, 1.57, 3.14, 4.71, and 6.28 rad/s. (Not all older individuals may be able to achieve the highest velocity – if not, the highest achieved angular velocity and associated torque will be used in all subsequent calculations.) The subject will perform 3-4 knee extensions at each velocity, with 2 minutes of rest allowed between each set of contractions. To eliminate artifacts, data will be "windowed" to isolate the isokinetic phase and smoothed using a 9 point weighted moving average filter using the manufacturer's software. The highest torque generated at each velocity will be used to calculate peak power at that velocity, after which the resulting power-velocity curve will be fit with a parabolic function to determine the subject's Pmax and Vmax (i.e., Y-

maximum and 2<sup>nd</sup> Y-intercept of fitted parabola, respectively) as previously described (30,33).

Measurement of perceived fatigue, physical function, and physical activity: Perceived fatigue and physical function will be assessed using PROMIS® Short Forms 8a and 20a, respectively, which are physical functioning questionnaires. Actual physical function will be quantified by the FIT Core using a suite of tests, i.e., usual gait speed, fast gait speed, Short Physical Performance Battery, 30 s chair stand performance, 6 min walk distance. Physical activity will be quantified using ActiGraph wGT3X-BT activity monitors (ActiGraph, Pensacola, FL). On Study Day 1, each participant will be given a fullycharged monitor and directed to wear the monitor on their right hip (superior to the iliac crest) for the next 7 days, removing it only when sleeping or during aquatic activities (i.e., bathing, swimming), and to complete a log of when the monitor is worn. On day 7, they will exchange the monitor for another, to be worn for the next 7 days. Upon return of the monitors, the data will be downloaded using the ActiLife 6 software, divided into 60 second epochs, and analyzed to quantify both total and bouted (i.e., >10 min duration) sedentary behavior, light physical activity, and moderate-to-vigorous physical activity (<100 counts/min, 100-2020, and >2020 counts/min, respectively). Total counts will also be recorded, since this may be more closely associated with the health benefits of physical activity (68). Results will be considered valid only if each monitor is worn for at least 10 hours/day over at least 4 days (including at least one weekend day) each week. Subsequently, the subject will perform an "all out" 50 contraction fatigue test (at 3.14 rad/s) to determine whether dietary NO3- influences fatigue resistance (i.e., increases average power) during repetitive, maximal activation. Finally, recovery of muscle function will be quantified by measuring restoration of torque during knee extensions performed periodically over the next 10 min.

## <u>Risks</u>

Beetroot Juice: Beetroot juice consumption or the consumption of the BRJ placebo may cause stool and/or urine to appear pink. This does NOT indicate bleeding. You may experience mild gastrointestinal distress (cramps, bloating) or diarrhea following ingestion of the BRJ. In rare cases there is a theoretical increased risk of upper GI cancers if a compound called "nitrosamine" is made from nitrates by the body. However, in large studies of many people followed up for many years, a fruit and vegetable-rich diet (where the acceptable daily intake of nitrates was exceeded several-fold) was not associated with any increase in cancer or mortality. The 2003 Joint Food and Agricultural Organization/World Health Organization Expert committee concluded that there was no evidence that nitrates are carcinogenic to humans.

Questionnaires: You may experience emotional discomfort when answering some questions in the health questionnaires. If any particular question makes you uncomfortable, you may discuss its importance and the need to answer it with the specially trained interviewer. You may choose not to answer any question with which you still feel uncomfortable.

*Needle Stick*: Slight pain, bruising or bleeding can occur. Rarely, infection can occur. Very infrequently, faintness may occur. To minimize the discomfort and risks associated with blood draw, only trained staff will collect blood samples.

*Exercise Test*: Your muscles may feel fatigued during the exercise test. You may also develop soreness in your muscles or joints. Very rarely, an exercise test, such as the neuromuscular function test, may be associated with serious complications including, but not limited to: fainting and disorders of the heart beat (too fast or too slow) which may require hospitalization; heart attack, stroke, or death; and muscle or joint pain. We will make every effort to minimize these rare risks by observing and monitoring during testing. However, no guarantees can be made. Emergency equipment and trained personnel are available to deal with any emergency.

*EKG:* some people may experience a skin rash but this usually goes away without treatment.

*Fit Core:* the risks for the Fit Core are described in that protocol (IRB study #1707550885).

Another risk of this study is the possible loss of confidentiality, which is minimal. Even though the risk is small, a link exists between your protected health information and your sample. In addition to the risks listed above, there may be some unknown or infrequent and unforeseeable risks associated with participation in this study. You will be informed in a timely manner of any new information, findings or changes to the way the research will be performed that might influence your willingness to continue your participation in this study.

## Mitigation of Risks

*Questionnaires*: Subjects may feel uncomfortable answering portions of the questionnaires. If so, they may discuss the importance of questions and the need to answer them with a member of the research team. They may choose not to answer any question with which they still feel uncomfortable.

Blood draw: Only trained staff will place IVs and collect blood samples

*Exercise test*: Every effort to minimize these rare risks by observing and monitoring during testing. Emergency equipment and trained personnel are available to deal with any emergency.

EKG: trained nurses will prepare the skin for the EKG and place the electrodes.

*Fit Core:* the mitigation of risks for the Fit Core are described in that protocol (IRB study #1707550885).

These instructions will be provided both verbally and in written form.

# 6.0 Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others

The following standard definitions will be used for this study:

## Adverse Event (AE)

Any untoward or unfavorable medical occurrence in a human study participant, including any abnormal sign (e.g. abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participants' involvement in the research, whether or not considered related to participation in the research.

## Serious Adverse Event (SAE)

Any AE that results is place the participant at immediate risk of death from the event as it occurred, or results in inpatient hospitalization, prolongation of existing hospitalization, persistent or significant disability/incapacity, congenital abnormalities or birth defects, or death.

### **Unanticipated Problem**

As Defined by DHHS 45 CFR part 46, any incident, experience, or outcome that meets all of the following criteria: 1) is unexpected, in terms of nature, severity, or frequency, given (a) the research procedures that are described in the protocol-related documents, such as the IRB-approved research protocol and informed consent document; and (b) the characteristics of the study population; 2) is related or possibly related to participation in the research (in this guidance document, possibly related means there is a reasonable possibility that the incident, experience, or outcome may have been caused by the procedures involved in the research); and 3) suggests that the research places participants or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized.

AEs will be graded according to the following scale:

- Mild: An experience that is transient, and requires no special treatment or intervention. The experience does not generally interfere with usual daily activities. This includes transient laboratory test alterations.
- Moderate: An experience that is alleviated with simple therapeutic treatments.
  The experience impacts usual daily activities. Includes laboratory test alterations indicating injury, but without long-term risk.
- Severe: An experience that requires therapeutic intervention. The experience interrupts usual daily activities. If hospitalization (or prolongation of hospitalization) is required for treatment it becomes an SAE.

Attribution of AEs and SAEs will be categorized as:

- *Not related*: The AE is clearly not related to the study procedures (i.e., another cause of the event is most plausible and/or a clinically plausible temporal sequence is inconsistent with the onset of the event).
- Possibly related: An event that follows a reasonable temporal sequence from the initiation of study procedures, but that could readily have been produced by a number of other factors.
- Related: The AE is clearly related to the study procedures.

Reporting of AEs, SAEs, and unanticipated problems will follow the guidelines of the IU Standard Operating Procedure for Reporting Unanticipated Problems and Noncompliance. Specifically, the following events will be reported promptly (i.e., within five business days) to the IRB:

- AEs (including SAEs) that are assessed by the PI or coinvestigators as (1) unexpected, (2) related or possibly related to participation, AND (3) suggests that the research places subject(s) or others at greater risk of harm than was previously known;
- Major protocol deviations that may, in the opinion of the PI, (1) impact subject safety, (2) affect the integrity of the data, OR (3) affect study participant' willingness to participate in the study;
- Noncompliance, which includes any action or activity associated with the conduct or oversight of the research that fails to comply with federal or state regulations, institutional policies governing human study participant research, or the requirements or determinations of the IRB.

Unanticipated problems that do not meet the criteria for prompt reporting will be reported at time of protocol renewal to ensure the IRB has a full understanding of the conduct of the research.

## 7.0 Study Withdrawal/Discontinuation

A participant may withdrawal from the study at any time verbally or by providing this request in writing as described in the informed consent document. As outlined in the consent document, if the participant/patient wishes to withdraw consent, the PI will:

- no longer use and take reasonable steps to destroy all blood/tissue samples and information
- not take back any research / analyses already completed

## 8.0 Statistical Considerations

Data analyses: The primary outcomes are muscle contractile function (i.e., Vmax and Pmax) and muscle cGMP concentration on day 1 and day 14, as separate outcomes.  $H_0$  is that they are not different while on BRJ w/  $NO_3^-$  versus on BRJ w/o  $NO_3^-$  and  $H_a$  is that they are greater while on BRJ w/  $NO_3^-$ . This hypothesis will be tested using a mixed model analysis of variance approach, with treatment ( $NO_3^-$ , placebo), sequence ( $NO_3^-$ -to-placebo, placebo-to- $NO_3^-$ ), and intervention period ( $1^{st}$ ,  $2^{nd}$ ) as fixed effects and subject as a random effect to account for repeated measurements. Carryover will be evaluated by first testing the effect of sequence, i.e., does the effect of treatment depend on

sequence. Assuming no carryover, analysis of treatment will proceed using both sets of data. The perceived fatigue, physical function (both obtained from the Fit Core protocol), and accelerometer data will be analyzed using functional and time series data analysis techniques. A two-sided P<0.05 will be considered significant. SAS 9.4 will be used for data analysis (SAS Institute, Cary, NC).

Sample size calculations: Samples size calculations were performed based on our preliminary data on  $NO_3$ -induced changes in Pmax in seven older study participant. Based on the observed effect size of 0.47 and assuming an  $\alpha$  of 0.05, N=10 would be required to achieve a power (1- $\beta$ ) of 0.80 and N=16 would be required to achieve a power of 0.90. To allow for screen failures and potential withdrawals, we will therefore enroll **100** study participants (to finish 16).

Potential limitations and alternatives considered: A possible limitation of the proposed study is the lack of direct demonstration that dietary  $NO_3^-$  results in an increase in NO specifically within muscle. This is because 1) the biological half-life of NO is extremely short (i.e., seconds), precluding measurement of its concentration in the muscle (or plasma) samples, and 2) existing stable isotopic methods only measure the rate of NO production via the NOS pathway. We will, however, measure changes in plasma  $NO_3^ /NO_2^-$  levels in response to dietary  $NO_3^-$ . We therefore do not consider the absence of direct measurements of muscle NO to be a significant limitation.

A potentially more important limitation to this research is the lack of pilot data for certain measurements. Thus, although we will have adequate power to detect increases in Vmax and Pmax), we cannot be assured that we will be able to detect differences in all of our endpoints. However, the proposed experiments would still provide the data needed to design a larger study that is adequately powered to detect changes in all variables.

### 9.0 Privacy/Confidentiality Issues

All study activities will be performed within areas respective of the participants' right to privacy.

Although there can be no absolute guarantee of confidentiality, every practical precaution will be taken.

Each study participant will be assigned a unique ID. Samples and information will be de-identified using this unique ID.

# 10.0 Follow-up and Record Retention

Study recruitment will be ongoing. The duration of the entire study is expected to be 24 months.

Any remaining blood samples will be de-identified and discarded. The de-identified data will be retained on computer files indefinitely. Hard copy study documents will be kept in a locked, file cabinet in a locked room. Electronic study information will be stored on a

specified, password-protected network that is backed up daily. Only the study team and the relevant personnel will have access. Files will be kept on site until 2 years after study completion, and then sent to a secure archiving facility. Files will be kept for 7 years after study completion per state law requirements.

#### 11.0 References

- 1. Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. *J Gerontol* 1994;49:M85–M94.
- 2. Kokkinos P, Myers J. Exercise and physical activity: clinical outcomes and applications. *Circulation* 2010;122:1637–1648.
- 3. Reid KF, Fielding RA. Skeletal muscle power: A critical determinant of physical functioning in older adults. *Exerc Sports Sci Rev* 2012:40:4-40. PMCID:PMC3245773.
- 4. Kaminski HJ, Andrade FH. Nitric oxide: biologic effects on muscle and role in muscle diseases. *Neuromuscular Disord* 2001;11:517-524.
- Maréchal G, Gaily P. Effects of nitric oxide on the contraction of skeletal muscle. *Cell Mol Life Sci* 1999;55:1088-1102.
- 6. Stamler JS, Meissner G. Physiology of nitric oxide in skeletal muscle. *Physiol Rev* 2001;81:209-237.
- 7. Suhr S, Gehlert S, Gau M, Bloch W. Skeletal muscle function during exercise fine-tuning of diverse subsystems by nitric oxide. *Int J Mol Sci* 2013;14:7109-7139. PMCID: PMC3645679.
- Lamb GD, Westerblad H. Acute effects of reactive oxygen and nitrogen species on the contractile function of skeletal muscle. *J Physiol* 2011;589:2119-2127. PMCID: PMC3098691
- 9. Evangelista AM, Rao VS, Filo AR, Marozkina NV, Doctor A, Jones D,. Gaston B, Guilford WH. Direct regulation of striated muscle myosins by nitric oxide and endogenous nitrosothiols. *PLOS One* 2010; 5:e11209. Doi:10.137/journal.pone.0011209. MCID: PMC2887846.
- 10. Francis SH, Busch JL, Corbin JD. cGMP-dependent protein kinases and cGMP phosphodiesterases in nitric oxide and cGMP action. *Pharmacol Rev* 2010;62:525-563. PMCID: PMC2964902.
- 11. Di Massimo C, Lo Presti R, Corbacelli C, Pompei A, Scarpelli P, De Amicis D, Caimi G, Tozzi Ciancarelli MG. Impairment of plasma nitric oxide availability in senescent healthy individuals: Apparent involvement of extracellular superoxide dismutase activity. *Clin Hemorheol Microcirc* 2006;35:231–237.
- 12. Di Massimo C, Scarpelli P, Di Lorenzo N, Caimi G, di Orio F, Ciancarelli MG. Impaired plasma nitric oxide availability and extracellular superoxide dismutase activity in healthy humans with advancing age. *Life Sci* 2006;78:1163-1167.
- 13. Nyberg M, Blackwell JR, Damsgaard R, Jones AM, Hellsten Y, Mortensen SP. Lifelong physical activity prevents an age-related reduction in arterial and skeletal muscle nitric oxide bioavailability in humans. *J Physiol* 2012;590:5361-5370. PMCID: PMC3515824.
- Nyakayiru J, Kouw IWK, Cermak NM, Senden JM, van Loon LJC, Verdijk LB. Sodium nitrate ingestion increases skeletal muscle nitrate content in humans. *J Appl Physiol* 2017 Jun 29:jap.01036.2016. doi: 10.1152/japplphysiol.01036.2016. [Epub ahead of print]

- 15. Richmonds CR, Boonyapisit K, Kusner LL, Kaminski HJ. Nitric oxide synthase in aging rat skeletal muscle. *Mech Aging Dev* 1999;109:177-189.
- Song W, Kwak H-B, Kim J-H, Lawler JM. Exercise training modulates the nitric oxide synthase profile in skeletal muscle from old rats. *J Gerontol A Biol Sci Med Sci* 2009;64A:540-549. PMCID: PMC2800810.
- 17. Scrage WE, Eisenach JH, Joyner MJ. Aging reduces nitric oxide- and prostaglandin-mediated vasodilation in exercise humans. *J Physiol* 2007;579:227-236. PMCID: PMC2075375.
- 18. Proctor DN, Parker BA. Vasodilation and vascular control in contracting muscle of the aging human. *Microcirculation* 2006;13:315-327.
- 19. Behnke BJ, Delp MD. Aging blunts the dynamics of vasodilation in isolated skeletal muscle resistance vessels. *J Appl Physiol* 2010;108:14-20. PMCID:PMC2885069.
- Hirai DM, Copp SW, Holdsworth CT, Ferguson SK, Musch TI, Poole DC. Effects of neuronal nitric oxide synthase inhibition on microvascular and contractile function in skeletal muscle of aged rats. *Am J Physiol Heart Circ Physiol* 2012;303:H1076-1084. PMCID:PMC3469646.
- 21. Heffernan KS, Chalé A, Hau C, Cloutier GJ, Phillips EM, Warner P, Nickerson H, Reid KF, Kuvin JT, Fielding RA. Systemic vascular function is associated with muscular power in older adults. *J Aging Res* 2012:2012:386387. Published online 2012 August 26. doi: 10.1155/2012/386387. PMCID:PMC3433136.
- 22. Lundberg JO, Weitzberg E, Gladwin MT. The nitrate—nitrite—nitric oxide pathway in physiology and therapeutics. *Nat Rev Drug Discov* 2008;7:156-167.
- 23. Lundberg JO, Weitzbefg E. NO generation from inorganic nitrate and nitrite: Role in physiology, nutrition, and therapeutics. *Arch Pharm Res* 2009;32:1119-1126.
- 24. Lundberg JO, Weitzberg E. NO-synthase independent NO generation in mammals. *Biochem Biophys Res Commun* 2010;396:39-45.
- 25. Gilchrist M, Winyard PG, Benjamin N. Dietary nitrate--good or bad? *Nitric Oxide* 2010;22:104-109.
- 26. Machha A, Schecter AN. Dietary nitrite and nitrate:a review of potential mechanisms of cardiovascular benefits. *Eur J Nutr* 2011;50:293-303. PMCID:PMC3489477.
- 27. Wagner DA, Schultz DS, Deen WM, Young VR, Tannenbaum SR. Metabolic fate of an oral dose of <sup>15</sup>N-labeled nitrate in humans: Effect of diet supplementation with ascorbic acid. *Cancer Res* 1983;43:1921-1925.
- 28. Siervo M, Stephan BCM, Feelisch M, Bluck LJC. Measurement of in vivo nitric oxide synthesis in humans using stable isotopic methods: a systematic review. *Free Radical Bio Med* 2011;51:795-804.
- 29. Piknova B, Park JW, Swanson KM, Dey S, Noguchi CT, Schechter AN. Skeletal muscle as an endogenous nitrate reservoir. *Nitric Oxide* 2015;47:10-16. PMCID: PMC4439352.
- 30. 34. Haider G, Folland JP. Nitrate supplementation enhances the contractile properties of human skeletal muscle. Med Sci Sports Exerc 2014; 46:2234-2243.
- 31. Whitfield J, Gamu D, Heigenhauser GJF, van Loon LJC, Spriet LL, Tupling AR, Holloway GP. Beetroot juice increases human muscle force without changing Ca<sup>2+</sup>-handling proteins. *Med Sci Sports Exerc.* 2017 May 15. doi: 10.1249/MSS.000000000001321. [Epub ahead of print]
- 32. Jones AM, Bailey SJ, Vanhatalo A. Dietary nitrate supplementation and exercise performance. *Sports Med* 2014;44:S35-S45.
- 33. Kelly J, Fulford J, Vanhatalo A, Blackwell JR, French O, Bailey SJ, Gilchrist M, Winyard PG, Jones AM. Effects of short-term dietary nitrate supplementation on blood

- pressure, O<sub>2</sub> uptake kinetics, and muscle and cognitive function in older adults. *Am J Physiol Regul Integr Comp Physiol* 2013;304:R73–R83.
- 34. Siervo M, Oggioni C, Jakovljevic DG, Trenell M, Mathers JC Houghton D, Celis-Morales C, Ashor AW, Ruddock A, Ranchordas M, Klonizakis M, Williams EA. Dietary nitrate does not affect physical activity or outcomes in healthy older adults in a randomized, cross-over trial. *Nutr Res* 2016; 36:1361-1369.
- 35. Shaltout HA, Eggebeen J, Marsh AP, Brubaker PH, Laurienti, PJ, Burdette JH, Basu S, Morgan A. Dos Santos PC, Norris JL, Morgan TM, Miller GD, Rejeski WJ, Hawfield AT, Diz DI, Becton JT, Kim-Shapiro DB, Kitzman DW. Effects of supervised exercise and dietary nitrate in older adults with controlled hypertension and/or heart failure with preserved ejection fraction. *Nitric Oxide* 2017; <a href="http://dx.doi.org/10.1016/j.niox.2017.05.005">http://dx.doi.org/10.1016/j.niox.2017.05.005</a>.
- 36. Justice JN, Johnson LC, DeVan AE, Cruickshank-Quinn C, Reisdorph N, Bassett CJ, Evans TD, Brooks FA, Bryan NS, Chonchol MB, Giordano T, McQueen MB, Seals DR. Improved motor and cognitive performance with sodium nitrite supplementation is related to small metabolite signatures: a pilot trial in middle-aged and older adults. *Aging* 2015; 7:1004-1021.
- 37. Coggan AR, Leibowitz JL, Kadkhodayan A, Thomas DT, Ramamurthy S, Anderson Spearie C, Waller S, Farmer M, Peterson LR. Effect of acute dietary nitrate intake on knee extensor speed and power in healthy men and women. *Nitric Oxide* 2015;48:16-21. PMCID: PMC4362985.
- 38. Rimer EG, Peterson LR, Coggan AR, Martin JC. Acute dietary nitrate supplementation increases maximal cycling power in athletes. Int J Sports Physiol Perf 2016; 11:715-720. PCMID: PMC4889556.
- 39. Kramer SJ, Baur DA, Spicer MT, Vukovich MD, Ormsbee MJ. The effect of six days of dietary nitrate supplementation on performance in trained CrossFit athletes. *J Int Soc Sports Nutr* 2016; 13:39. DOI: 10.1186/s12970-016-0150-y.
- 40. Ferguson AK, Hirai DM, Copp SW, Holdsworth CT, Allen JD, Jones AM, Musch TI, Poole DC. Impact of dietary nitrate supplementation via beetroot juice on exercising muscle vascular control in rats. *J Physiol* 2013;591:547-555. PMCID: PMC3577528.
- 41. Hernández A, Schiffer TA, Ivarsson N, Cheng AJ, Bruton JD, Lundberg JO, Weitzberg E, Westerblad H. Dietary nitrate increases tetanic [Ca<sup>2+</sup>]<sub>1</sub> and contractile force in mouse fast-twitch muscle. *J Physiol* 2012;590:3575-3583. PMCID: PMC3547271.
- 42. Larsson L, Grimby G, Karlsson J. Muscle strength and speed of movement in relation to age and muscle morphology. *J Appl Physiol* 1979;46:451-456.
- 43. Lexell J. Human aging, muscle mass, and fiber type composition. *J Gerontol A Biol Sci Med Sci* 1995;50A:11-16.
- 44. Lee WS, Cheung WH, Qin L, Tang N, Leung KS. Age-associated decrease of type IIA/B human skeletal muscle fibers. *Clin Orthop Relat Res* 2006;450:231-237.
- 45. Marzani B, Felzani G, Bellomo RG, Vecchiet J, Marzatico F. Human skeletal muscle aging: ROS-mediated alterations in rectus abdominis and vastus lateralis muscles. *Exp Gerontol* 2005;40:959-965.
- 46. Coggan AR, Spina RJ, Rogers MA, King DS, Brown M, Nemeth PM, Holloszy JO. Histochemical and enzymatic comparison of the gastrocnemius muscle of young and elderly men and women. *J Geront* 1992;47:B71-B76.
- 47. Frontera WR, Reid KF, Phillips EM, Krivickas LS, Hughes VA, Roubenoff R, Fielding RA. Muscle fiber size and function in elderly humans: a longitudinal study. *J Appl Physiol* 2008;105:637-642. PMCID: PMC2519941.

- 48. Verdijk LB, Dirks ML, Snijders T, Prompers JJ, Beelen M, Jonkers RA, Thijssen DH, Hopman MT, Van Loon LJ. Reduced satellite cell numbers with spinal cord injury and aging in humans. *Med Sci Sports* Exerc 2012;44:2322-2330.
- 49. Doria E, Buonocore D, Focarelli A, Marzatico F. Relationship between human aging muscle and oxidative system pathway. *Oxid Med Cell Longev* 2012;2012:803257. Doi: 10.1155/2012/830257. Epub 2012 May 17.
- 50. Crandall LA, Leake AS, Loevenhart AS, Muehlberger CW. Acquired tolerance to and cross tolerance between the nitrous and nitric acid esters and sodium nitrite in man. *J Pharmacol Exp Therapeut* 1931;41:103-119.
- 51. Dejam A, Hunter CJ, Tremonti C, Pluta RM, Hon YY, Grimes G, Partovi K, Plelletier MM, Oldfield EH, Cannon RO, Schechter AN, Gladwin MT. Nitrite infusion in humans and nonhuman primates. Endocrine effects, pharmacokinetics, and tolerance formation. *Circulation* 2007;116:1821-1831.
- 52. Coggan AR, Leibowitz JL, Anderson Spearie C, Kadkhodayan A, Thomas DP, Ramamurthy S, Mahmood K, Park S, Waller S, Farmer M, Peterson LR. Acute dietary nitrate intake improves muscle contractile function in patients with heart failure: a double-blind, placebo-controlled, randomized trial. *Circ Heart Fail* 2015;8:914-920. PMCID: PMC4573847.
- 53. Katz SD, Khan T, Zeballos GA, Mathew L, Potharlanka P, Knecht M, Whelan J. Decreased activity of the L-arginine-nitric oxide metabolic pathway in patients with congestive heart failure. *Circulation*. 1999; 99:2113-2117.
- 54. Miller GD, Marsh AP, Dove RW, Beavers D, Presley T, Helms C, Bechtold E, King BS, Kim-Shapiro D. Plasma nitrate and nitrite are increased by a high-nitrate supplement but not by high-nitrate foods in older adults. *Nutr Res* 2012;32:160-168. PMCID: PMC3319660.
- 55. Wylie LJ, Kelly J, Bailey SJ, Blackwell JR, Skiba PF, Winyard PG, Jeukendrup AE, Vanhatalo A, Jones AM. Beetroot juice and exercise: pharmacodynamic and doseresponse relationships. *J Appl Physiol* 2013;115:325-336.
- 56. Olin AC, Aldenbratt A, Ekman A, Ljungkvist G, Jungersten L, Alving K, Torén K. Increased nitric oxide in exhaled air after intake of a nitrate-rich meal. *Resp Med* 2001:95:153-158.
- 57. Vints AM, Oostveen E, Eeckhaut G, Smolders M, De Backer WA. Time-dependent effect of nitrate-rich meals on exhaled nitric oxide in healthy subjects. *Chest* 2005;128;2465-70.
- 58. Gilchrist M, Winyard PG, Aizawa K, Anning C, Shore A, Benjamin N. Effect of dietary nitrate on blood pressure, endothelial function, and insulin sensitivity in type 2 diabetes. *Free Radic Bio Med* 2013; 60:89-97.
- 59. Cermak NM, Hansen D, Kouw IW, van Dikk JW, Blackwell JR, Jones AM, Gibala MJ, va Loon LJ. A single dose of sodium nitrate does not improve oral glucose tolerance in patients with type 2 diabetes. *Nutr Res* 2015; 35:674-680.
- 60. Ashor AW, Chowdhury S, Oggioni C, Qadur O, Brandt K, Ishaq A, Mathers JC, Saretzki G, Siervo M. Inorganic nitrate supplementation in young and old obese adults does not affect acute glucose and insulin responses but lowers oxidative stress. *J Nutr* 2016; 146:2224-2232.
- 61. Gregory CM, Bickel CS. Recruitment patterns in human skeletal muscle during electrical stimulation. *Phys Ther* 2005;85:358-364.
- 62. Derave W, Taes Y. Beware of the pickle: health effects of nitrate intake. *J Appl Physiol* 2009;107:1677; author reply 1678.

- 63. Hord NG, Tang Y, Bryan NS. Food sources of nitrates and nitrites: the physiologic context for potential health benefits. *Am J Clin Nutr* 2009;90:1-10.
- 64. Griesenbeck JS, Steck MD, Huber JC Jr, Sharkey JR, Rene AA, Brender JD. Development of estimates of dietary nitrates, nitrites, and nitrosamines for use with the Short Willet Food Frequency Questionnaire. *Nutr J.* 2009;8:16. doi:10.1186/1475-2891-8-16. PMCID: PMC2669451.
- 65. Jungersten L, Edlund A, Petersson AS, Wennmalm A. Plasma nitrate as an index of nitric oxide formation in man: analyses of kinetics and confounding factors. *Clin Physiol* 1996:16:369-379.
- 66. Govoni M, Jansson EA, Weitzberg E, Lundberg JO. The increase in plasma nitrite after a dietary nitrate load is markedly attenuated by an antibacterial mouthwash. *Nitric Oxide* 2008;19:333-337.